CLINICAL TRIAL: NCT00422656
Title: A Phase II Study of Perifosine in Patients With Relapsed/Refractory Waldenstrom's Macroglobulinemia
Brief Title: Perifosine in Patients With Relapsed/Refractory Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-077
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Results first posted 2012-02-16 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: relapsed Waldenstrom's Macroglobulinemia; refractory Waldenstrom's Macroglobulinemia; WM; perifosine
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — perifosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perifosine (Experimental): Patients receive oral perifosine (150 mg) daily each cycle. Cycle duration is 28 days. After cycle 2, response is assessed and patients with stable or responding disease can continue for another 4 cycles or until disease progression (PD). Protocol treatment duration is 6 cycles but patients may receive perifosine maintenance per investigator discretion in absence of PD.
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine
  Other Names: KRX-0401

SUMMARY:
Waldenström's Macroglobulinemia (lymphoplasmacytic lymphoma, WM) remains incurable with limited therapeutic options and notably absent FDA approved therapy with any WM indication. Therefore, there is a need to identify new therapeutic agents for WM patients both in the upfront and relapsed/refractory setting. The purpose of this research study is to assess the efficacy of perifosine in patients with relapsed or refractory WM.

DETAILED DESCRIPTION:
Perifosine is a drug that in particular inhibits Akt thought to be important for initiation and progression of malignancies, specifically in lymphomas. In laboratory experiments of WM and lymphoma cell lines, perifosine has shown to have cytotoxic and anti-proliferative activity as a single agent. This drug has been used in clinical research studies of other types of cancers including soft tissue sarcomas, head and neck cancers and prostate cancer. This study uses a two-stage design to evaluate efficacy of perifosine based on overall response (OR). The null and alternative OR rates are 20% and 40%. If 4 or more patients enrolled in the stage one cohort (n=17 patients) achieve OR than accrual will proceed to stage two (n=20 patients). If fewer than 10 ORs are observed then the regimen will be considered ineffective.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must have received prior therapy for their WM and have relapsed or refractory WM. Any number of prior therapies is acceptable
* Measurable disease, defined as presence of immunoglobulin M paraprotein with a minimum IgM level of equal to or greater than 2 times the ULN and over 10% of lymphoplasmacytic cells in bone marrow
* ECOG Performance Status 0,1, or 2
* Laboratory values as described in the protocol
* Life expectancy of greater than 12 weeks

Exclusion Criteria:

* Uncontrolled infection
* Other active malignancies
* CNS involvement
* Cytotoxic chemotherapy less than 3 weeks, or biologic therapy less than 2 weeks, or corticosteroids less than 2 weeks prior to registration.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational
* Pregnant or nursing women
* Known to be HIV positive
* Radiation therapy less than 2 weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ghobrial IM, Roccaro A, Hong F, Weller E, Rubin N, Leduc R, Rourke M, Chuma S, Sacco A, Jia X, Azab F, Azab AK, Rodig S, Warren D, Harris B, Varticovski L, Sportelli P, Leleu X, Anderson KC, Richardson PG. Clinical and translational studies of a phase II trial of the novel oral Akt inhibitor perifosine in relapsed or relapsed/refractory Waldenstrom's macroglobulinemia. Clin Cancer Res. 2010 Feb 1;16(3):1033-41. doi: 10.1158/1078-0432.CCR-09-1837. Epub 2010 Jan 26. PMID 20103671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2006 through November 2007, patients enrolled from the Dana-Farber Cancer Institute in Boston, MA as well as at the Community Hospital of Monterey Peninsula in Monterey, CA.
Period: Overall Study
Arm/Group | Perifosine
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Perifosine
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR) Rate
Description: OR rate is the percentage of patients achieving Complete Response (CR), Partial Response (PR) or Minimal Response (MR) during treatment based on criteria from the 2nd International Workshop on WM. (Weber D, Treon S, et al. Seminars in Oncology 2003). CR: Disappearance of serum monoclonal IgM protein (IgM M-protein) by immunofixation; no histologic evidence of bone marrow (BM) involvement, resolution of any adenopathy/organomegaly (confirmed by CT scan); PR: At least 50% reduction of IgM M-protein and at least 50% decrease in adenopathy/organomegaly on physical examination or on CT scan; and MR: At least 25% but less than 50% reduction of IgM M-protein by protein electrophoresis. Patients must have no new symptoms or signs of active disease.
Time Frame: Disease was assessed every cycle for the first 12 months and every 3 months thereafter. The median duration of treatment with perifosine was 5.6 months (range, 1.8- 21.5+).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Perifosine
Number analyzed (Participants) | 37
percentage of patients | 38 [25 to 53]

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP estimated using the Kaplan-Meier method is defined as the time from registration to disease progression (PD) based on criteria from the 2nd International Workshop on WM. (Weber D, Treon S, et al. Seminars in Oncology 2003) Patients without PD are censored at time of last disease assessment. PD: At least 25% increase in serum monoclonal IgM protein by electrophoresis confirmed with a second measurement at least 2 weeks apart, or progression of clinically significant findings due to disease (i.e., anemia, thrombocytopenia, leucopenia, bulky adenopathy/organomegaly) or symptoms (unexplained recurrent fever of at least 38.4oC, drenching night sweats, at least 10% body weight less, or hyperviscosity, neuropathy, symptomatic cryoglobulinemia, or amyloidosis) attributable to WM.
Time Frame: Disease was assessed every cycle for the first 12 months and every 3 months thereafter. Median follow-up time was 19.5 months and range up to 24 months.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Perifosine
Number analyzed (Participants) | 37
months | 12.6 [10.2 to 22.7]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS estimated using the Kaplan-Meier method is defined as the time from registration to death from any cause or disease progression (PD) based on criteria from the 2nd International Workshop on WM. (Weber D, Treon S, et al. Seminars in Oncology 2003) Patients alive without PD are censored at time of last disease assessment. PD: At least 25% increase in serum monoclonal IgM protein by electrophoresis confirmed with a second measurement at least 2 weeks apart, or progression of clinically significant findings due to disease (i.e., anemia, thrombocytopenia, leucopenia, bulky adenopathy/organomegaly) or symptoms (unexplained recurrent fever of at least 38.4oC, drenching night sweats, at least 10% body weight less, or hyperviscosity, neuropathy, symptomatic cryoglobulinemia, or amyloidosis) attributable to WM.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Perifosine
Number analyzed (Participants) | 37
months | 12.6 [10.2 to 22.7]

4. Secondary Outcome: Treatment-Related Grade 3-4 Adverse Event Rate
Description: The percentage of patients experiencing treatment-related grade 3-4 adverse events based on CTCAEv3 as reported on case report forms.
Time Frame: Adverse events were collected every cycle on treatment.The median treatment duration was 5.6 months (range, 1.8-21.5+).
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Perifosine
Number analyzed (Participants) | 37
percentage of patients | 35 [22 to 50]

ADVERSE EVENTS:
Time Frame: Adverse events were collected every cycle on treatment.The median treatment duration was 5.6 months (range, 1.8-21.5+).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Arm/Group | Perifosine
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 14/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perifosine (N=37)
Hemoglobin (Blood and lymphatic system disorders) | 1
Vision-blurred (Eye disorders) | 1
Eye, pain (Eye disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Infection Gr0-2 neut, bronchus (Infections and infestations) | 1
Leukocytes (Investigations) | 5
Neutrophils (Investigations) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Gastritis/Dyspepsia (Gastrointestinal disorders) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perifosine (N=37)
Tinnitus (Ear and labyrinth disorders) | 2
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 26
Palpitations (Cardiac disorders) | 2
Hearing-other (Ear and labyrinth disorders) | 1
Vision-blurred (Eye disorders) | 8
Ocular-other (Eye disorders) | 2
Eye, pain (Eye disorders) | 4
Constipation (Gastrointestinal disorders) | 13
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 30
Distention/bloating, abdominal (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 10
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 25
Oral cavity, hemorrhage (Gastrointestinal disorders) | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 2
Abdomen, pain (Gastrointestinal disorders) | 3
Stomach, pain (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 27
Fever w/o neutropenia (General disorders) | 3
Rigors/chills (General disorders) | 1
Edema limb (General disorders) | 2
Pain-other (General disorders) | 2
Flu-like syndrome (General disorders) | 3
Infection Gr0-2 neut, middle ear (Infections and infestations) | 1
Infection-other (Infections and infestations) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Haptoglobin (Investigations) | 2
Leukocytes (Investigations) | 20
Lymphopenia (Investigations) | 4
Neutrophils (Investigations) | 19
Platelets (Investigations) | 3
Weight gain (Investigations) | 2
Weight loss (Investigations) | 10
INR (Investigations) | 1
Alkaline phosphatase (Investigations) | 5
ALT, SGPT (Investigations) | 3
AST, SGOT (Investigations) | 4
Bilirubin (Investigations) | 7
Creatinine (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 24
Alkalosis (Metabolism and nutrition disorders) | 1
Bicarbonate (Metabolism and nutrition disorders) | 14
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 17
Hyperglycemia (Metabolism and nutrition disorders) | 28
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 19
Hyponatremia (Metabolism and nutrition disorders) | 6
Hyperuricemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 6
Bone, pain (Musculoskeletal and connective tissue disorders) | 3
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 5
Joint, pain (Musculoskeletal and connective tissue disorders) | 6
Taste disturbance (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Extrapyramidal movement (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 9
Seizure (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 9
Sinus, pain (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Psychosis (Psychiatric disorders) | 1
Libido (Psychiatric disorders) | 2
Hemoglobinuria (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 1
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, airway-bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Odor (patient odor) (Skin and subcutaneous tissue disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Skin-other (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No